CLINICAL TRIAL: NCT03829904
Title: The Effect of Traditional Chinese Medicine VGH-BPH1 on Patients With Benign Prostatic Hyperplasia: A Double-blinded Randomized Placebo-controlled Cross-over Study
Brief Title: The Effect of Traditional Chinese Medicine on Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-01-019C
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Traditional Chinese medicine
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Starch

STUDY DESIGN:
Intervention Model Description: 40 participants will be recruited from Division of Urology in a Medical Center. They will be randomizedly allocated into treatment and control groups, each including 20 participants. After eight weeks of taking, there is a two weeks of drug wash-out period. And then two groups will be switched for another eight weeks. The study duration is totally 18 weeks.
Who Masked: Participant, Investigator
Masking Description: Placebo is manufactured to have the same appearance with VGH-BPH1, after that VGH-BPH1 and placebo will be coded as package A and B by the manufacturer and the codes will only be revealed after the study ends. Therefore, patients and investigators will not know which package is VGH-BPH1 or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VGH-BPH1 group (Experimental): VGH-BPH1 includes Ji Sheng Shen Qi Wan 2.5g, Sangpiaoxiao powder 1.0g, Wuyao 0.3g, Yizhiren 0.3g, Danshen 0.3g, Yinyanghuo 0.3g, Fupenzi 0.1g, Huangbo 0.25g and Zhimu 0.25g, three times per day, each serving a small packet of 5.3 grams of concentrated granules.
  Interventions: Drug: VGH-BPH1
- Control group (Placebo Comparator): Placebo includes corn starch plus caramel coloring, and added 1/100 VGH-BHP1 compound, three times per day, each serving a small packet of 5.3 grams of concentrated granules.
  Interventions: Drug: Placebo (Corn starch pill manufactured to mimic VGH-BPH1)

INTERVENTIONS:
Drug: VGH-BPH1 — A scientific Chinese granule powder
  Arms: VGH-BPH1 group
Drug: Placebo (Corn starch pill manufactured to mimic VGH-BPH1) — Corn starch pill manufactured to mimic VGH-BPH1
  Arms: Control group

SUMMARY:
This randomized, double-blinded, placebo-controlled, crossover clinical trial aims to investigate the effect of VGH-BPH1, a scientific Chinese medicine powder prescription, on patients with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is an enlargement of the prostate gland due to progressive hyperplasia of the stromal and glandular cells.

The aim of this study is to evaluate the efficacy of traditional Chinese medicine (VGH-BPH1) in treating patients with BPH, by using the experimental BPH-1 powder, including Ji Sheng Shen Qi Wan and Sangpiaoxiao powder as the main prescription, and adding Wuyao, Yizhiren, Danshen, Yinyanghuo, Fupenzi, Huangbo and Zhimu as auxiliary ingredients, to form a 5gm per pack. This study is designed as a double-blinded randomized placebo-controlled cross-over trial to provide experimental evidence and feasibility of traditional Chinese medicine VGH-BPH1 in the treatment of BPH, and to analyze the syndrome pattern of Chinese medicinal prescriptions for subgroups of BPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with benign prostatic hyperplasia by a urologist
* Have been treated with conventional first-line western medicine for more than three months
* Patients with moderate to severe benign prostatic hyperplasia (IPSS score >12 points)
* Participate voluntarily in the study

Exclusion Criteria:

* At the same time, use other Chinese herbal medicines or alternative medicine (including drugs and acupuncture) for more than one month.
* Syphilis, gonorrhea and other sexually transmitted diseases or urinary tract infections
* Urinary tract stones, prostate cancer, bladder cancer or acute and chronic renal failure
* Congenital abnormalities such as bladder neck fibrosis, interstitial cystitis or urethral stricture
* A history of genital trauma or surgery affecting the muscle or nervous system
* Patients with upper urinary tract obstruction, renal edema, etc. affecting renal function
* Unable to sign a consent form or unable to communicate with researchers

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male patients who have been diagnosed with benign prostatic hyperplasia
Enrollment: 23 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
International prostate symptom score (IPSS) | Change from Baseline IPSS at eight weeks, ten weeks, eighteen weeks
  To measure the severity of lower urinary tract symptoms. Each item is scored 0-5, yielding a total between 0-35.
Aging Male Symptoms score (AMS) | Change from Baseline AMS at eight weeks, ten weeks, eighteen weeks
  To evaluate health-related quality of life in aging men. Each item is scored 1-5, yielding a total between 17-85.

SECONDARY OUTCOMES:
Constitution in Chinese Medicine Questionnaire (CCMQ) | Change from Baseline CCMQ at eight weeks, ten weeks, eighteen weeks
  It has 60 items measuring the 9 body constitution types: gentleness, Qi-deficiency, Yang-deficiency, Yin-deficiency, phlegm-wetness, wetness-heat, blood-stasis, Qi-depression, and special diathesis.
Post-voiding residual urine | Change from Baseline post-voiding residual urine at eight weeks, ten weeks, eighteen weeks
  To measure and compare the amount of urine left in the bladder after urination before and after treatment.
International index of erectile function (IIEF) | Change from Baseline IIEF at eight weeks, ten weeks, eighteen weeks
  To evaluate male sexual function over the past 6 months. Each item is scored 1-5, yielding a total between 5-25.
Maximum flow rate (Qmax) and Average flow rate (Qave） | Change from Baseline Qmax and Qave at eight weeks, ten weeks, eighteen weeks
  To determine peak urine flow rate and average urine flow rate. They are calculated by ml/sec.
Voided volume (VV) | Change from Baseline VV at eight weeks, ten weeks, eighteen weeks
  To calculate the amount of urine (ml)
Voiding time and time to maximum flow | Change from Baseline Voiding time and time to maximum flow at eight weeks, ten weeks, eighteen weeks
  To calculate the length of time it takes to empty bladder completely and the peak urine flow time (sec)

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Jang Hwang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nickel JC. The overlapping lower urinary tract symptoms of benign prostatic hyperplasia and prostatitis. Curr Opin Urol. 2006 Jan;16(1):5-10. doi: 10.1097/01.mou.0000193365.46081.cd. PMID 16385194
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Barqawi AB, Myers JB, O'Donnell C, Crawford ED. The effect of alpha-blocker and 5alpha-reductase inhibitor intake on sexual health in men with lower urinary tract symptoms. BJU Int. 2007 Oct;100(4):853-7. doi: 10.1111/j.1464-410X.2007.07092.x. Epub 2007 Jul 23. PMID 17662074
- [Background] Miner M, Rosenberg MT, Perelman MA. Treatment of lower urinary tract symptoms in benign prostatic hyperplasia and its impact on sexual function. Clin Ther. 2006 Jan;28(1):13-25. doi: 10.1016/j.clinthera.2006.01.004. PMID 16490576
- [Background] Jung JH, Jae SU, Kam SC, Hyun JS. Correlation between Lower Urinary Tract Symptoms (LUTS) and sexual function in benign prostatic hyperplasia: impact of treatment of LUTS on sexual function. J Sex Med. 2009 Aug;6(8):2299-304. doi: 10.1111/j.1743-6109.2009.01324.x. Epub 2009 Jun 2. PMID 19493292
- [Background] Sarma AV, Wei JT. Clinical practice. Benign prostatic hyperplasia and lower urinary tract symptoms. N Engl J Med. 2012 Jul 19;367(3):248-57. doi: 10.1056/NEJMcp1106637. No abstract available. PMID 22808960
- [Background] Pasko P, Rodacki T, Domagala-Rodacka R, Owczarek D. Interactions between medications employed in treating benign prostatic hyperplasia and food - A short review. Biomed Pharmacother. 2016 Oct;83:1141-1145. doi: 10.1016/j.biopha.2016.08.021. Epub 2016 Aug 20. PMID 27551761
- [Background] Tacklind J, Fink HA, Macdonald R, Rutks I, Wilt TJ. Finasteride for benign prostatic hyperplasia. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD006015. doi: 10.1002/14651858.CD006015.pub3. PMID 20927745
- [Background] Corona G, Tirabassi G, Santi D, Maseroli E, Gacci M, Dicuio M, Sforza A, Mannucci E, Maggi M. Sexual dysfunction in subjects treated with inhibitors of 5alpha-reductase for benign prostatic hyperplasia: a comprehensive review and meta-analysis. Andrology. 2017 Jul;5(4):671-678. doi: 10.1111/andr.12353. Epub 2017 Apr 28. PMID 28453908
- [Background] Li MK, Garcia L, Patron N, Moh LC, Sundram M, Leungwattanakij S, Pripatnanont C, Cheng C, Chi-Wai M, Loi-Cheong N. An Asian multinational prospective observational registry of patients with benign prostatic hyperplasia, with a focus on comorbidities, lower urinary tract symptoms and sexual function. BJU Int. 2008 Jan;101(2):197-202. doi: 10.1111/j.1464-410X.2007.07320.x. Epub 2007 Nov 13. PMID 18005205
- [Background] Wilt TJ, Ishani A, Stark G, MacDonald R, Lau J, Mulrow C. Saw palmetto extracts for treatment of benign prostatic hyperplasia: a systematic review. JAMA. 1998 Nov 11;280(18):1604-9. doi: 10.1001/jama.280.18.1604. PMID 9820264
- [Background] Pagano E, Laudato M, Griffo M, Capasso R. Phytotherapy of benign prostatic hyperplasia. A minireview. Phytother Res. 2014 Jul;28(7):949-55. doi: 10.1002/ptr.5084. PMID 25165780
- [Background] Keehn A, Lowe FC. Complementary and alternative medications for benign prostatic hyperplasia. Can J Urol. 2015 Oct;22 Suppl 1:18-23. PMID 26497340
- [Background] Ho CC, Singam P, Hong GE, Zainuddin ZM. Male sexual dysfunction in Asia. Asian J Androl. 2011 Jul;13(4):537-42. doi: 10.1038/aja.2010.135. Epub 2011 Jun 6. PMID 21643001
- [Background] Yagi H, Sato R, Nishio K, Arai G, Soh S, Okada H. Clinical efficacy and tolerability of two Japanese traditional herbal medicines, Hachimi-jio-gan and Gosha-jinki-gan, for lower urinary tract symptoms with cold sensitivity. J Tradit Complement Med. 2015 Apr 18;5(4):258-61. doi: 10.1016/j.jtcme.2015.03.010. eCollection 2015 Oct. PMID 26587398
- [Background] Chen F, Li HL, Li YH, Tan YF, Zhang JQ. Quantitative analysis of the major constituents in Chinese medicinal preparation SuoQuan formulae by ultra fast high performance liquid chromatography/quadrupole tandem mass spectrometry. Chem Cent J. 2013 Jul 30;7(1):131. doi: 10.1186/1752-153X-7-131. PMID 23899222
- [Background] Ge FH, Ma XP, Ma JF, Bi CQ, Chen TL, Zhang XD, Xiao X. Qualitative and Quantitative Characterization of Monosaccharide Components of Salvia miltiorrhiza, Liguspyragine Hydrochloride, and Glucose Injection. J Anal Methods Chem. 2017;2017:9245620. doi: 10.1155/2017/9245620. Epub 2017 Apr 11. PMID 28487814
- [Background] Chen F, Li L, Tian DD. Salvia miltiorrhiza Roots against Cardiovascular Disease: Consideration of Herb-Drug Interactions. Biomed Res Int. 2017;2017:9868694. doi: 10.1155/2017/9868694. Epub 2017 Apr 3. PMID 28473993
- [Background] Bonesi M, Loizzo MR, Acquaviva R, Malfa GA, Aiello F, Tundis R. Anti-inflammatory and Antioxidant Agents from Salvia Genus (Lamiaceae): An Assessment of the Current State of Knowledge. Antiinflamm Antiallergy Agents Med Chem. 2017;16(2):70-86. doi: 10.2174/1871523016666170502121419. PMID 28464779
- [Background] Jiang G, Liu J, Ren B, Zhang L, Owusu L, Liu L, Zhang J, Tang Y, Li W. Anti-tumor and chemosensitization effects of Cryptotanshinone extracted from Salvia miltiorrhiza Bge. on ovarian cancer cells in vitro. J Ethnopharmacol. 2017 Jun 9;205:33-40. doi: 10.1016/j.jep.2017.04.026. Epub 2017 Apr 27. PMID 28456578
- [Background] Deng Y, Long L, Wang K, Zhou J, Zeng L, He L, Gong Q. Icariside II, a Broad-Spectrum Anti-cancer Agent, Reverses Beta-Amyloid-Induced Cognitive Impairment through Reducing Inflammation and Apoptosis in Rats. Front Pharmacol. 2017 Feb 2;8:39. doi: 10.3389/fphar.2017.00039. eCollection 2017. PMID 28210222
- [Background] Mo ZT, Li WN, Zhai YR, Gao SY. The effects of icariin on the expression of HIF-1alpha, HSP-60 and HSP-70 in PC12 cells suffered from oxygen-glucose deprivation-induced injury. Pharm Biol. 2017 Dec;55(1):848-852. doi: 10.1080/13880209.2017.1281968. PMID 28140748
- [Background] Li XA, Ho YS, Chen L, Hsiao WL. The Protective Effects of Icariin against the Homocysteine-Induced Neurotoxicity in the Primary Embryonic Cultures of Rat Cortical Neurons. Molecules. 2016 Nov 22;21(11):1557. doi: 10.3390/molecules21111557. PMID 27879670
- [Background] Chen KK, Chiu JH. Effect of Epimedium brevicornum Maxim extract on elicitation of penile erection in the rat. Urology. 2006 Mar;67(3):631-5. doi: 10.1016/j.urology.2005.09.051. PMID 16527595
- [Background] Chang CM, Wu PC, Chiang JH, Wei YH, Chen FP, Chen TJ, Pan TL, Yen HR, Chang HH. Integrative therapy decreases the risk of lupus nephritis in patients with systemic lupus erythematosus: A population-based retrospective cohort study. J Ethnopharmacol. 2017 Jan 20;196:201-212. doi: 10.1016/j.jep.2016.12.016. Epub 2016 Dec 12. PMID 27974236